CLINICAL TRIAL: NCT04249336
Title: Immediate And Sustained Treatment Response Of Commercially Available BioMin F, Colgate Sensitive Pro-Relief And Sensodyne Rapid Action Dentifrices In Dentin Hypersensitivity - "A Randomized Clinical Trial"
Brief Title: Clinical Efficacy Of BioMin F, Colgate Sensitive Pro-Relief And Sensodyne Rapid Action Dentifrices In DH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Syed Jaffar Abbas Zaidi, Principal investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRS4072
Record Dates: First submitted 2019-09-26; First posted 2020-01-30 (Actual); Results first posted 2021-05-11 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-04

CONDITIONS: Dentin Hypersensitivity
Keywords: Dentine hypersensitivity; Dentine Sensitivity; Oral dentifrices; Bio-active glasses
MeSH Terms: conditions — Dentin Sensitivity | interventions — strontium acetate; Sodium Fluoride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Statistician will be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- BioMin F Dentifrices (Experimental): Participants will be instructed to dose a dry toothbrush with a full strip of dentifrices and to brush teeth for 1 minute twice daily.
  Interventions: Drug: Fluoro-Calcium-Phospho-Silicate based dentifrices
- Colgate Sensitive Pro relief Trade Mark Dentifrices (Active Comparator): Participants will be instructed to dose a dry toothbrush with a full strip of dentifrices and to brush teeth for 1 minute twice daily.
  Interventions: Drug: 8% Arginine based dentifrices
- Sensodyne Rapid Action Trade Mark Dentifrices (Active Comparator): Participants will be instructed to dose a dry toothbrush with a full strip of dentifrices and to brush teeth for 1 minute twice daily.
  Interventions: Drug: 8% Strontium Acetate
- Colgate Total Trade Mark (Placebo Comparator): Participants will be instructed to dose a dry toothbrush with a full strip of dentifrices and to brush teeth for 1 minute twice daily.
  Interventions: Drug: Sodium Fluoride

INTERVENTIONS:
Drug: Fluoro-Calcium-Phospho-Silicate based dentifrices — Bio-Active glass based formulation
  Other Names: BioMin F
  Arms: BioMin F Dentifrices
Drug: 8% Arginine based dentifrices — Tubular occluding formulation
  Other Names: Colgate Sensitive Pro-Relief TM
  Arms: Colgate Sensitive Pro relief Trade Mark Dentifrices
Drug: 8% Strontium Acetate — Tubular occluding formulation
  Other Names: Sensodyne Rapid ActionTM
  Arms: Sensodyne Rapid Action Trade Mark Dentifrices
Drug: Sodium Fluoride — No claim of relieving Dentin Hypersensitivity
  Other Names: Colgate Total TM
  Arms: Colgate Total Trade Mark

SUMMARY:
This will be multi-centered, triple blinded, randomized, four parallel treatments assigned study to compare clinical efficacy of commercially available dentifrices with placebo for immediate and sustained relief from Dentin Hypersensitivity after short term use.

Condition or disease: Dentin hypersensitivity Intervention/Treatment: Product 1; Fluoro-Calcium-Phospho-silicate based BioMin F Product 2; Pro-Argin formula based Colgate Sensitive Pro-Relief Product 3; Strontium Acetate based Sensodyne Rapid Action Product 4; Sodium Fluoride based Colgate Total

DETAILED DESCRIPTION:
It is a randomized controlled clinical trial with non invasive topical intervention in 140 adult patients of 18 to 60 years age, that will be selected randomly after screening and diagnosis of dentin hypersensitivity, in dental Out Patient Department of Periodontology. Written informed consent will be obtained. Participants will be allocated randomly into four equal study arms for parallel treatment assignment with dentifrices named BioMin F, Colgate Sensitive Pro-Relief Trade Mark,Sensodyne rapid action Trade Mark and Colgate Total Trade Mark dentifrices. Colgate total Trade Mark dentifrices does not claim pain relief in Dentin Hypersensitivity. Interim efficacy will be assessed immediately after topical application on sensitive teeth, in one minute, after 5 minutes, on day three and week 4 respectively. Dentin hypersensitivity will be tested with mechanical stimulus, evaporative air blast stimulus and water jet stimulus. It will be measured on Visual Analogue Scale and Schiff cold air sensitivity scale (SCASS). Statistical analysis will be done using ANOVA in Statistical Package for Social Sciences software 21.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with at least two teeth sensitive to cold, touch and air blow stimulus
* Sensitive teeth anterior to molars either due to erosions or abrasions with or without associated gingival recession
* Teeth with Linear Visual Analogue Scale (VAS) score of ≥ 4 and code 2 of Schiff Cold Air Sensitivity Scale on screening.

Exclusion Criteria:

* Subjects with worst pain response at 100mm on VAS.(Visual Analog Scale)
* Teeth with orthodontic or prosthetic appliances, Caries, restorations or cracks
* Localized or generalized gingivitis or pulpitis with heavy calculus
* Periodontal surgery in the preceding three months
* Patients using any desensitizing tooth paste or mouth wash up to six weeks before study and taking drugs like anti-inflammatory, sedatives, tranquilizers, analgesics in routine.
* Pregnant or breastfeeding females.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2019-09-27 (Actual); Primary Completion 2021-01-16 (Actual); Study Completion 2021-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Syed Jaffar Abbas Zaidi, Study Director — Dow University of Health Sciences
Locations (1):
- Dr Syed Jaffar Abbas Zaidi, Karachi, Sindh, Pakistan

REFERENCES:
- [Background] Hall C, Mason S, Cooke J. Exploratory randomised controlled clinical study to evaluate the comparative efficacy of two occluding toothpastes - a 5% calcium sodium phosphosilicate toothpaste and an 8% arginine/calcium carbonate toothpaste - for the longer-term relief of dentine hypersensitivity. J Dent. 2017 May;60:36-43. doi: 10.1016/j.jdent.2017.02.009. Epub 2017 Feb 20. PMID 28219674
- [Background] Ashwini S, Swatika K, Kamala DN. Comparative Evaluation of Desensitizing Efficacy of Dentifrice Containing 5% Fluoro Calcium Phosphosilicate versus 5% Calcium Sodium Phosphosilicate: A Randomized Controlled Clinical Trial. Contemp Clin Dent. 2018 Jul-Sep;9(3):330-336. doi: 10.4103/ccd.ccd_735_17. PMID 30166822
- [Derived] Arshad S, Zaidi SJA, Farooqui WA. Comparative efficacy of BioMin-F, Colgate Sensitive Pro-relief and Sensodyne Rapid Action in relieving dentin hypersensitivity: a randomized controlled trial. BMC Oral Health. 2021 Oct 6;21(1):498. doi: 10.1186/s12903-021-01864-x. PMID 34615511

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited and enrolled based on self reported sensitivity in teeth followed by clinical diagnosis of dentin hypersensitivity using Air blast stimulus response on SCHIFF Air Blast Sensitivity Scale at Department of Periodontology, Dr. Ishrat-ul-Ibad Khan Institute of Oral Health Sciences, DUHS, Karachi between September 2019 to December 2020. The first Participant was enrolled in September 27, 2019 and last participant was enrolled in October 2020.
Pre-assignment Details: Of 380 assessed participants of self reported sensitivity in teeth, 140 met inclusion criteria and were randomized to treatment.
Groups:
- Colgate Sensitive Pro Relief: Participants received Colgate Sensitive Pro relief Trademark Dentifrices and instructed to brush their teeth with a full strip of dentifrices on a dry toothbrush for 1 minute twice daily for 4 weeks.
  Colgate Sensitive Pro relief Trade Mark Dentifrices : 8% Arginine and calcium carbonate, tubular occluding formulation
- BioMin F: Participants received BioMin F Dentifrices and instructed to brush their teeth with a full strip of dentifrices on a dry toothbrush for 1 minute twice daily for 4 weeks.
  BioMin F Dentifrices : Fluoro-Calcium-Phospho-Silicate, Bio-Active glass based tubular occluding formulation
- Sensodyne Rapid Action: Participants received Sensodyne Rapid Action dentifrices and instructed to brush their teeth with a full strip of dentifrices on a dry toothbrush for 1 minute twice daily for 4 weeks.
  Sensodyne Rapid Action Trademark Dentifrices : 8% Strontium Acetate with tubular occluding formulation.
- Colgate Total: Participants received Colgate Total dentifrices and instructed to brush their teeth with a full strip of dentifrices on a dry toothbrush for 1 minute twice daily for 4 weeks.
  Colgate Total Trademark Dentifrices : Sodium Fluoride with no claim of relieving Dentin Hypersensitivity
Period: Overall Study
Arm/Group | Colgate Sensitive Pro Relief | BioMin F | Sensodyne Rapid Action | Colgate Total
Started | 35 | 35 | 35 | 35
Per Protocol Population Day 3 | 32 | 32 | 32 | 32
Per Protocol Population Week 4 | 33 | 35 | 33 | 34
Completed (Out of 35 participants per group, 32 completed the 4-week clinical trial after lost to follow up and statistically analyzed for primary outcome measure.) | 32 | 32 | 32 | 32
Not Completed | 3 | 3 | 3 | 3
Not completed — Lost to Follow-up | 3 | 3 | 3 | 3

BASELINE CHARACTERISTICS:
Population: 35 individuals per treatment group were recruited and enrolled in the study after clinical diagnosis of dentin hypersensitivity using air blast stimulus and SCHIFF cold air sensitivity scale. These participants were tested again for dentin hypersensitivity using mechanical stimulus and Visual Analogue Scale. After lost to follow up, statistical analysis was performed for 32 participants per group with baseline SCHIFF scale score of ≥2 and visual Analogue Scale score of ≥4.
Groups:
- BioMin F Dentifrices: Participants were instructed to dose a dry toothbrush with a full strip of dentifrices and to brush teeth for 1 minute twice daily.
  Fluoro-Calcium-Phospho-Silicate based dentifrices: Bio-Active glass based formulation
- Colgate Sensitive Pro Relief Trademark Dentifrices: Participants were instructed to dose a dry toothbrush with a full strip of dentifrices and to brush teeth for 1 minute twice daily.
  8% Arginine based dentifrices: Tubular occluding formulation
- Sensodyne Rapid Action Trademark Dentifrices: Participants were instructed to dose a dry toothbrush with a full strip of dentifrices and to brush teeth for 1 minute twice daily.
  8% Strontium Acetate: Tubular occluding formulation
- Colgate Total Trademark: Participants were instructed to dose a dry toothbrush with a full strip of dentifrices and to brush teeth for 1 minute twice daily.
  Sodium Fluoride: No claim of relieving Dentin Hypersensitivity
- Total: Total of all reporting groups
Arm/Group | BioMin F Dentifrices | Colgate Sensitive Pro Relief Trademark Dentifrices | Sensodyne Rapid Action Trademark Dentifrices | Colgate Total Trademark | Total
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 128
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.23 (8.77) | 34.40 (8.43) | 35.63 (9.55) | 34.14 (9.08) | 34.10 (8.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 21 | 17 | 20 | 80
  Male | 10 | 11 | 15 | 12 | 48
Race (NIH/OMB) [Count of Participants; unit: Participants] — Asian (Pakistani) population was studied in 4 week clinical trial.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
    Asian | 32 | 32 | 32 | 32 | 128
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 0 | 0
    White | 0 | 0 | 0 | 0 | 0
    More than one race | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Summary of the baseline SCHIFF cold air sensitivity scale for air blast stimulus response [Mean (Standard Deviation); unit: scores on a scale] — SCHIFF cold air sensitivity scale was used to measure the intensity of pain due to dentin hypersensitivity using air blast stimulus. Patients' response of pain was assessed by the doctor according to following score criteria; "0" for no response of pain, "1" for pain response but no request of discontinuity of stimulus, "2" for pain response with request of discontinuity of stimulus, "3" for Immediate pain response for discontinuity of stimulus Population: Total lost to follow up was 12 out of 140 enrolled participants. Lost to follow up per group was 3 out of 35. Statistical analysis was performed for 32 participants per group.
  scores on a scale | 2.46 (0.50) | 2.46 (0.50) | 2.46 (0.50) | 2.46 (0.50) | 2.46 (0.50)
Summary of the baseline Visual Analog scale for Mechanical and Water jet stimulus response [Mean (Standard Deviation); unit: scores on a scale] — Visual Analogue Scale was used to measure the intensity of pain due to dentin hypersensitivity using mechanical stimulus and water jet stimulus. Patient's response of pain was assessed on vertical line of 0 to 10cm by asking him to move finger on the line and stop it where he felt pain. Scoring criteria for each cm was, 0cm for no pain with score 0, 1-3cm for mild pain with scores 1,2 and 3, 4-6cm for moderate pain with scores 4,5 and 6, 7-9cm for severe pain with scores 7,8 and 9 and 10cm for worst imaginable pain with score10. Population: Out of 35 participants per group, 20 participants responded on Visual Analogue Scale for DH in 4-week trial.
  scores on a scale
    Mechanical hypersensitivity baseline score: number analyzed (Participants) | 20 | 20 | 20 | 20 | 80
    Mechanical hypersensitivity baseline score | 6.75 (0.91) | 6.70 (1.03) | 6.70 (1.17) | 6.70 (1.03) | 6.71 (1.02)
    Water Jet hypersensitivity baseline score: number analyzed (Participants) | 20 | 20 | 20 | 20 | 80
    Water Jet hypersensitivity baseline score | 6.70 (0.80) | 6.18 (2.23) | 6.75 (0.91) | 6.48 (1.69) | 6.52 (1.54)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Mean Score of Pain Response From Baseline on Schiff Cold Air Sensitivity Scale Using Air Blast Stimulus
Description: SCHIFF cold air sensitivity scale was used to measure the intensity of pain due to dentin hypersensitivity using air blast stimulus. Patients' response of pain was assessed by the doctor according to following score range from; "0"(no response of pain), "1" (pain response but no request of discontinuity of stimulus), "2"(pain response with request of discontinuity of stimulus), "3"(Immediate pain response for discontinuity of stimulus). Percent change in mean scores = ( one minute score-Baseline score) / Baseline score
Time Frame: (Base line to 1 minute) (Base line to 5 minutes)(Base line to day 3)(Base line to week 4)
Population: 35 individuals per treatment group were recruited and enrolled in the study after clinical diagnosis of dentin hypersensitivity using air blast stimulus and SCHIFF cold air sensitivity scale. These participants were tested again for dentin hypersensitivity using mechanical stimulus and Visual Analogue Scale. After lost to follow up, statistical analysis was performed for 32 participants per group with baseline SCHIFF scale score of ≥2.
Measure: Mean (Standard Deviation); unit: percentage of change in mean scores
Arm/Group | BioMin F | Colgate Sensitive Pro Relief | Sensodyne Rapid Action | Colgate Total
Number analyzed (Participants) | 32 | 32 | 32 | 32
percentage of change in mean scores
  1- minute | 18 (21) | 45 (24) | 37 (27) | 15 (22)
  5-minutes | 27 (22) | 56 (25) | 51 (28) | 19 (21)
  Day-3 | 22 (22) | 24 (21) | 25 (21) | 10 (18)
  Week-4 | 58 (26) | 55 (24) | 45 (25) | 22 (24)
Statistical Analysis 1: Comparison: BioMin F vs Colgate Total; It was calculated that 140 participants randomized in a 1:1:1:1 fashion between the four arms would have at least 80 % power to detect a difference of 0.20 mean scores between four treatments from baseline to week 4. Sample size was determined using PAS V.11, two independent sample t-test with 95% confidence interval; Test type: Superiority; p < 0.05, ANOVA — Threshold for statistical significance was p <0.05; Mean Difference (Net) = 36 — Treatment difference in percent = BioMin F- Colgate Total
Statistical Analysis 2: Comparison: Colgate Sensitive Pro Relief vs Colgate Total; Test type: Superiority; p < 0.05, ANOVA — Threshold P<0.05; Mean Difference (Net) = 33 — Treatment difference in percent = Colgate Sensitive Pro relief - Colgate Total
Statistical Analysis 3: Comparison: Sensodyne Rapid Action vs Colgate Total; Test type: Superiority; p < 0.05, ANOVA — Threshold for statistical significance was p <0.05; Mean Difference (Net) = 23 — Treatment difference in percent = Sensodyne Rapid Action - Colgate Total

2. Secondary Outcome: Percent Change in Mean Scores of Pain Response From Baseline on Visual Analog Scale Using Mechanical Stimulus
Description: Visual Analogue Scale was used to measure the intensity of pain due to dentin hypersensitivity using mechanical stimulus. Patient's response of pain was assessed on vertical line of 0 to 10cm by asking him to move finger on the line and stop it where he felt pain. Score range from; 0 (no pain at 0cm), 1(mild pain at 1cm), 2(mild pain at 2cm), 3(mild pain at 3cm), 4(moderate pain at 4cm), 5(moderate pain at 5cm), 6(moderate pain at 6cm), 7(severe pain at 7cm), 8(severe pain at 8cm), 9(severe pain at 9cm),10(worst imaginable pain at 10cm). Percent change in mean scores = (one minute score-Baseline score) / Baseline score
Time Frame: (Base line to 1 minute) (Base line to 5 minutes)(Base line to day 3)(Base line to week 4)
Population: 35 individuals per treatment group were recruited and enrolled in the study after clinical diagnosis of dentin hypersensitivity using air blast stimulus and SCHIFF cold air sensitivity scale. These participants were tested again for dentin hypersensitivity using mechanical stimulus and Visual Analogue Scale. Statistical analysis was performed for 20 participants out of 32 per group with visual Analogue Scale score of ≥4.
Measure: Mean (Standard Deviation); unit: percentage of change in mean scores
Arm/Group | BioMin F | Colgate Sensitive Pro Relief | Sensodyne Rapid Action | Colgate Total
Number analyzed (Participants) | 20 | 20 | 20 | 20
percentage of change in mean scores
  1-minute | 25 (22) | 56 (27) | 46 (26) | 16 (13)
  5-minutes | 27 (23) | 61 (26) | 51 (27) | 20 (13)
  Day-3 | 28 (15) | 38 (20) | 32 (20) | 18 (12)
  Week-4 | 59 (27) | 66 (27) | 57 (27) | 27 (16)
Statistical Analysis 1: Comparison: BioMin F vs Colgate Total; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.05, ANCOVA — Threshold for statistical significance was p <0.05; Mean Difference (Net) = 32 — Treatment difference in percent = BioMin F- Colgate Total
Statistical Analysis 2: Comparison: Colgate Sensitive Pro Relief vs Colgate Total; Test type: Superiority; p < 0.05, ANOVA — Threshold for statistical significance was p <0.05; Mean Difference (Net) = 39 — Treatment difference in percent = Colgate Sensitive Pro relief - Colgate Total
Statistical Analysis 3: Comparison: Sensodyne Rapid Action vs Colgate Total; Test type: Superiority; p < 0.05, ANOVA — Threshold for statistical significance was p <0.05; Mean Difference (Net) = 30 — Treatment difference in percent = Sensodyne Rapid Action - Colgate Total

3. Secondary Outcome: Percent Change in Mean Scores of Pain Response From Baseline on Visual Analog Scale Using Water Jet Stimulus
Description: Visual Analogue Scale was used to measure the intensity of pain due to dentin hypersensitivity using Water Jet Stimulus. Patient's response of pain was assessed on vertical line of 0 to 10cm by asking him to move finger on the line and stop it where he felt pain. Score range from; 0 (no pain at 0cm), 1(mild pain at 1cm), 2(mild pain at 2cm), 3(mild pain at 3cm), 4(moderate pain at 4cm), 5(moderate pain at 5cm), 6(moderate pain at 6cm), 7(severe pain at 7cm), 8(severe pain at 8cm), 9(severe pain at 9cm),10(worst imaginable pain at 10cm). Percent change in mean scores = (one minute score-Baseline score) / Baseline score
Time Frame: (Base line to 1 minute) (Base line to 5 minutes)(Base line to day 3)(Base line to week 4)
Population: 35 individuals per treatment group were recruited and enrolled in the study after clinical diagnosis of dentin hypersensitivity using air blast stimulus and SCHIFF cold air sensitivity scale. These participants were tested again for dentin hypersensitivity using water jet stimulus and Visual Analogue Scale. Statistical analysis was performed for 20 participants out of 32 with Visual Analogue Scale score of ≥4.
Measure: Mean (Standard Deviation); unit: percentage of change in mean scores
Arm/Group | BioMin F | Colgate Sensitive Pro Relief | Sensodyne Rapid Action | Colgate Total
Number analyzed (Participants) | 20 | 20 | 20 | 20
percentage of change in mean scores
  1-minute | 22 (21) | 52 (26) | 46 (25) | 18 (15)
  5-minutes | 27 (22) | 56 (25) | 52 (24) | 21 (17)
  Day-3 | 30 (29) | 34 (22) | 32 (21) | 18 (16)
  Week-4 | 67 (25) | 57 (23) | 55 (22) | 29 (20)
Statistical Analysis 1: Comparison: BioMin F vs Colgate Total; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.05, ANCOVA — Threshold for statistical significance was p <0.05; Median Difference (Net) = 36 — Treatment difference in percent = BioMin F- Colgate Total
Statistical Analysis 2: Comparison: Colgate Sensitive Pro Relief vs Colgate Total; Test type: Superiority; p < 0.05, ANOVA — Threshold for statistical significance was p <0.05; Mean Difference (Net) = 28 — Treatment difference in percent = Colgate Sensitive Pro relief - Colgate Total
Statistical Analysis 3: Comparison: Sensodyne Rapid Action vs Colgate Total; Test type: Superiority; p < 0.05, ANOVA — Threshold for statistical significance was p <0.05; Mean Difference (Net) = 25 — Treatment difference in percent = Sensodyne Rapid Action - Colgate Total

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | BioMin F Dentifrices | Colgate Sensitive Pro Relief Trade Mark Dentifrices | Sensodyne Rapid Action Trade Mark Dentifrices | Colgate Total Trade Mark
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35 | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35 | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35 | 0/35 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-09-07): https://cdn.clinicaltrials.gov/large-docs/36/NCT04249336/Prot_SAP_000.pdf
  • Informed Consent Form (2019-09-07): https://cdn.clinicaltrials.gov/large-docs/36/NCT04249336/ICF_001.pdf